CLINICAL TRIAL: NCT00131560
Title: A Phase II, Open-label, Multicenter Study to Evaluate the Safety, Tolerability, and Biological Activity of Single and Repeated Doses of Autologous T Cells Transduced With VRX496 in HIV-Positive Subjects
Brief Title: Safety and Efficacy of T Cell Genetic Immunotherapy for HIV
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: VIRxSYS Corporation (Industry)
Responsible Party: Tessio Rebello/ Vice President Clinical Affairs, VIRxSYS Corporation
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VRX496-USA-05-002
Record Dates: First submitted 2005-08-16; First posted 2005-08-18 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: HIV Infection
Keywords: HIV, gene therapy, leukapheresis, autologous CD4 T cell, lentivector
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Other)
  Interventions: Genetic: VRX496-Modified Autologous T cells

INTERVENTIONS:
Genetic: VRX496-Modified Autologous T cells — Genetic: Anti-HIV antisense

SUMMARY:
This study uses autologous (one's own) CD4 T cells modified with a viral vector expressing a genetic antisense targeting HIV, this vector is called VRX496. Study treatment is by intravenous infusion of vector modified cells and infusions will be provided every other week for a total of 4 or 8 doses. These modified cells, once infused, may provide immune support and are not destroyed by HIV, and thus may delay or reverse HIV disease progression. The study will enroll up to 40 male and female HIV-positive subjects in up to 8 centers. Subjects will be 18 years of age and over who have failed or are intolerant to at least one triple combination of antiretroviral drugs. Subjects must have a viral load between 5,000 and 200,000 copies/ml and a CD4+ count of ≥150, be in good health and have no evidence of active opportunistic infection, heart disease, or bleeding disorders. Subjects must not be on corticosteroids, immunomodulating agents or hydroxyurea. Subjects must not have received an AIDS vaccine or any investigational gene therapy product at any time. Females must not be pregnant or breastfeeding.

DETAILED DESCRIPTION:
VIRxSYS has concluded a 6-month Phase 1/2 clinical study under an IND of the vector VRX496 in HIV-positive subjects who have failed at least two HAART regimens. HAART typically consists of a triple "cocktail" of drugs. Although these cocktails have been successful in reducing viral loads and restoring immune function, they do not represent a cure. There are also concerns about adverse effects associated with long-term usage of HAART. Specifically, a variety of metabolic disorders including HIV-associated lipodystrophy, central adiposity, dyslipidaemia, hyperlipidaemia, hyperglycemia, and insulin resistance have been reported as resulting from HAART. These reactions, combined with often complex and cumbersome dosing regimens, can have an adverse effect on patient-subject adherence to therapy. Furthermore, poor adherence has led to increased rates of HIV resistance, resulting in viral strains that have reduced sensitivity to the drugs. Importantly, in the Phase 1/2 clinical trial conducted by VIRxSYS, there were no reported toxicities associated with the product.

Gene therapy for HIV-1 infection has been proposed as an alternative to antiretroviral drug regimens. A number of different genetic vectors with antiviral payloads have been utilized to combat HIV-1, including antisense RNA, transdominant proteins, ribozymes, RNA decoys, single chain antibodies, and RNAi (RNA-interference. Antisense RNA targeted to wt-HIV RNA offers a significant advantage over several other genetic antiviral approaches because it is not a protein and thus not immunogenic and because the size of the payload prevents virus escape mutants, such as occurs with the use of RNAi.

In this Phase 2 protocol, 6 subjects will be staggered for infusion by at least 2 weeks. The first group of 3 subjects will receive 4 infusions (4-dose cohort). If no dose limiting toxicities (DLT) are observed, the second group of 3 subjects, (i.e. subjects 4, 5 and 6) will continue with 8 infusions (8-dose cohort). Safety visits are scheduled 1 week after infusion and monthly for the first 6 months and at 9 months following the last infusion.

After safety has been evaluated, and in order to explore biological activity, additional subjects (6-10 evaluable subjects) will be entered into each cohort. Follow-up visits are scheduled 1 week after infusion and monthly for the first 6 months and at 9 months following the last infusion.

The effect of a single bolus will also be examined in a third cohort. The single bolus infusion will consist of the following cell doses: approximately 10 billion, 20 billion, and 30 billion, respectively. Subjects will be allotted to the respective cell dose groups according to the order in which they are enrolled. Three to 5 subjects will be allotted to the lower cell dose group and followed for safety for 4 weeks. After safety is evaluated, the next group (3 to 5 subjects) will be allotted to the next higher cell dose group and followed for safety for 4 weeks. If the intermediate cell dose group is determined to be safe, an additional 3 to 5 subjects will be allotted to the highest cell dose group. All subjects will be followed for safety at biweekly intervals for the first 4 weeks and thereafter at monthly intervals up to 6 months and then at 9 months.

The study has concluded it's 9-month active phase. Subjects are currently in a 15-year Long Term Follow-up Phase of the study.

In keeping with the recently released Guidance on Monitoring For Delayed Adverse Events, that states that for the first 5 years all subjects should undergo monitoring of vector sequences every 6 months, subjects will visit the clinic at a maximum of 6 months intervals for a blood test evaluating persistence of vector sequences.

Therefore for the first 5 years, subjects will have 6 months visits for safety assessment. For years 6 to 15, subjects will be contacted by phone or mail. At these contacts, subjects will be asked about their health status.

ELIGIBILITY:
Inclusion Criteria:

* Sero-positive for infection with HIV and failed, or be intolerant to, at least one triple combination of antiretroviral agent
* If on antiretroviral therapy, subject must be willing to continue on current antiretroviral therapy; or if discontinues antiretroviral therapy must have a wash-out period of 6 weeks prior to screening; or if not on antiretroviral therapy must be willing to remain off antiretroviral therapy for the duration of the study (i.e. up to 1 year)
* Male or female, 18 years of age and older
* Karnofsky Performance score of 80 or higher
* Stable HIV viral load between 5,000 and 200,000 copies/mL at the time of screening. Stable will be defined as a variation of less than 0.5 log10 in the 3 months prior to screening while on a stable regimen or no therapy
* CD4 T cell count equal to or greater than 150 cells per μL at the time of screening
* A body weight greater than 50 Kg
* Adequate venous access and no other contraindications for leukapheresis
* Subject must be willing to comply with study-mandated evaluations

Exclusion Criteria:

* A history of any type of cancer or malignancy, with the exception of (successfully) treated basal cell or squamous cell carcinoma of the skin
* A history or any features on physical examination indicative of cardiac disease or hemodynamic instability
* Any history or any features on physical examination indicative of a bleeding diathesis
* Previous treatment with any HIV experimental vaccine or any gene therapy products
* A positive signal for VSV-G antibodies and/or VSV-G DNA in the blood at screening
* Any of the following lab results:

  * Hemoglobin: <10 (males); <9.5 (females) g/dL
  * Absolute neutrophil count: < 1000/μL
  * Platelet count: <100,000/mm3
  * Serum creatinine: > 1.5 mg/dL (133µ mol/L)
  * AST or ALT: > 2.5 times the upper limit of normal
  * Total serum bilirubin: > 1.5 times the upper limit of normal
  * Proteinuria: 2+ on urine dipstick
* Subjects must not be breastfeeding, be pregnant, or unwilling to use acceptable methods of birth control
* Subjects must not be on chronic oral corticosteroids within 30 days of screening - (if subjects are prescribed a brief course of oral corticosteroids the use should be limited to less than 1 week), hydroxyurea, or immunomodulating agents (e.g., IL 2, interferon-gamma, granulocyte colony stimulating factors, etc.) within 30-days of screening or foreseeably need any of these within the study period
* Subjects must not be using aspirin, dipyridamole, warfarin or any other medication likely to affect platelet function or other aspects of blood coagulation during the period when leukapheresis is scheduled
* Subjects must not suffer from active drug or alcohol dependence or abuse, to an extent that, in the opinion of the investigator, would interfere with their ability to comply with study requirements
* Any serious illnesses or acute opportunistic infection
* Any other illness or condition which in the opinion of the investigator would exclude the subject from the study
* Subjects unable or unwilling to give written informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2005-07; Primary Completion 2008-11 (Actual); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Change in viral load | 1 Year
Change in CD4 counts | 1 Year
Safety | 15 Years

SECONDARY OUTCOMES:
Immune function | 1 Year
AIDS related illness | 1 Year
Persistence of vector modified cells | 15 Years

CONTACTS AND LOCATIONS:
Overall Officials: Tessio Rebello, PhD, Study Director — VIRxSYS Corporation
Locations (5):
- United States (5):
  - Stanford AIDS Clinical Trials Unit, Palo Alto, California
  - CIRCLE Medical, LLC, Norwalk, Connecticut
  - Steinhart Medical Associates, Miami, Florida
  - University of Kentucky, Lexington, Kentucky
  - Jacobi Medical Center, The Bronx, New York

REFERENCES:
- [Background] Manilla P, Rebello T, Afable C, Lu X, Slepushkin V, Humeau LM, Schonely K, Ni Y, Binder GK, Levine BL, MacGregor RR, June CH, Dropulic B. Regulatory considerations for novel gene therapy products: a review of the process leading to the first clinical lentiviral vector. Hum Gene Ther. 2005 Jan;16(1):17-25. doi: 10.1089/hum.2005.16.17. PMID 15703485
- [Background] Ni Y, Sun S, Oparaocha I, Humeau L, Davis B, Cohen R, Binder G, Chang YN, Slepushkin V, Dropulic B. Generation of a packaging cell line for prolonged large-scale production of high-titer HIV-1-based lentiviral vector. J Gene Med. 2005 Jun;7(6):818-34. doi: 10.1002/jgm.726. PMID 15693055
- [Background] Lu X, Humeau L, Slepushkin V, Binder G, Yu Q, Slepushkina T, Chen Z, Merling R, Davis B, Chang YN, Dropulic B. Safe two-plasmid production for the first clinical lentivirus vector that achieves >99% transduction in primary cells using a one-step protocol. J Gene Med. 2004 Sep;6(9):963-73. doi: 10.1002/jgm.593. PMID 15352069
- [Background] Lu X, Yu Q, Binder GK, Chen Z, Slepushkina T, Rossi J, Dropulic B. Antisense-mediated inhibition of human immunodeficiency virus (HIV) replication by use of an HIV type 1-based vector results in severely attenuated mutants incapable of developing resistance. J Virol. 2004 Jul;78(13):7079-88. doi: 10.1128/JVI.78.13.7079-7088.2004. PMID 15194784
- [Background] Humeau LM, Binder GK, Lu X, Slepushkin V, Merling R, Echeagaray P, Pereira M, Slepushkina T, Barnett S, Dropulic LK, Carroll R, Levine BL, June CH, Dropulic B. Efficient lentiviral vector-mediated control of HIV-1 replication in CD4 lymphocytes from diverse HIV+ infected patients grouped according to CD4 count and viral load. Mol Ther. 2004 Jun;9(6):902-13. doi: 10.1016/j.ymthe.2004.03.005. PMID 15194057
- See also: VIRxSYS Corporation website — http://www.virxsys.com